CLINICAL TRIAL: NCT03166930
Title: Evaluation of a Spasticity Management Program for People With Multiple Sclerosis
Acronym: STC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B2507-R; I01RX002507 (NIH)
Record Dates: First submitted 2017-05-19; First posted 2017-05-25 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Muscle Spasticity; Muscle Stretching Exercises
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two exercise programs. Participants will not be masked regarding which group they are in, but they will not be told which group is considered standard of care and which is the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spasticity Take Control (Experimental): Participants will attend two 2-hour classes via video teleconference (online), one week apart, consisting of education and a stretching program for spasticity management.
  Interventions: Behavioral: Spasticity Take Control
- Stretching for People with MS: An Illustrated Manual (Active Comparator): Participants will attend two 2-hour classes via video teleconference (online), one week apart, consisting of education and exercises for spasticity management.
  Interventions: Behavioral: Stretching for People with MS: An Illustrated Manual

INTERVENTIONS:
Behavioral: Spasticity Take Control — Participants will attend two 2-hour classes via video teleconference (online), one week apart, consisting of education and a stretching program for spasticity management.
  Arms: Spasticity Take Control
Behavioral: Stretching for People with MS: An Illustrated Manual — Participants will attend two 2-hour classes via video teleconference (online), one week apart, consisting of education and exercises for spasticity management from the manual.
  Arms: Stretching for People with MS: An Illustrated Manual

SUMMARY:
This study will examine the impacts of two different methods of managing MS-related spasticity of the lower limbs. Both interventions will be presented via video teleconference in group classes consisting of exercises to reduce spasticity.

DETAILED DESCRIPTION:
Now online since COVID-19

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of definite MS by 2010 updated McDonald Criteria
* Age 18 or older
* Able to walk 25 feet with any assistive devices (Patient Determined Disease Steps 0-6)
* Fluent in written and spoken English, as materials are not validated in languages other than English.
* Presence of self-reported lower extremity spasticity that is interfering with daily activities or sleep, using the this definition: Have spasticity in your legs with unusual tightening of muscles that feels like leg stiffness, jumping of the legs, a repetitive bouncing of the foot, muscle cramping in the legs, or the legs going out tight and straight or drawing up.
* All women that meet the above criteria
* Only Veteran men that meet the above criteria

Exclusion Criteria:

* Any uncontrolled medical or mental condition that would limit participation or completion of the study
* Any self-reported musculoskeletal or neurological condition other than MS that is known to cause spasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Impact of spasticity, measured by the Multiple Sclerosis Spasticity Scale-88 | One month post-intervention
  Impact of spasticity will be measured using the Multiple Sclerosis Spasticity Scale-88 at one month post intervention.

SECONDARY OUTCOMES:
Severity of spasticity, measured by the Numeric Rating Scale for Spasticity | One month post-intervention
  Severity of spasticity will be measured using the Numeric Rating Scale for Spasticity at one month post intervention.
Fatigue, measured by the Modified Fatigue Impact Scale | One month post-intervention
  Fatigue will be measured using the Modified Fatigue Impact Scale at one month post intervention.
Sleep quality and quantity, measured by the Pittsburge Sleep Quality Index | One month post-intervention
  Sleep quality and quantity will be measured using Pittsburgh Sleep Quality Index at one month post intervention.
Impact on day-to-day life, measured by the Multiple Sclerosis Impact Scale-29 | One month post-intervention
  Impact on day-to-day life, measured by the Multiple Sclerosis Impact Scale-29 at one month post intervention.
PROMIS Item Bank v1.0 - Emotional Distress - Depression-Short Form 8a | One month post-intervention
  Emotional Distress - Depression will be measured using PROMIS Item Bank v1.0 - Emotional Distress - Depression-Short Form 8a at one month post intervention.
Impact on multiple sclerosis on walking, measured by the Multiple Sclerosis Walking Scale-12 | One month post-intervention
  Impact on multiple sclerosis on walking, measured by the Multiple Sclerosis Walking Scale-12 at one month post intervention.
Walking measured by the Timed 25 Foot Walk | One month post-intervention
  Walking will be measured using the Timed 25 Foot Walk at one month post intervention, only if visit is in person.
Walking and turning measured by the Timed Up and Go | One month post-intervention
  Walking and turning measured by the Timed Up and Go will be measured at one month post intervention, only if visit is in person.

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda L. Hugos, PT MS, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hugos CL, Cameron MH. MS Spasticity: Take Control (STC) for ambulatory adults: protocol for a randomized controlled trial. BMC Neurol. 2020 Oct 7;20(1):368. doi: 10.1186/s12883-020-01902-1. PMID 33028236